CLINICAL TRIAL: NCT01709227
Title: Early Renal Replacement Therapy vs. Furosemide for Neonates With Oliguria After Cardiopulmonary Bypass
Brief Title: Peritoneal Dialysis vs Furosemide for Acute Kidney Injury After Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1730
Record Dates: First submitted 2012-09-20; First posted 2012-10-18 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; AKI; cardiopulmonary bypass
MeSH Terms: conditions — Acute Kidney Injury | interventions — Furosemide; Peritoneal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Furosemide (Experimental): Patients randomized to the furosemide arm will be given 1 mg/kg intravenously every 6 hours for 2 doses and then as directed by CICU attending to augment urine output. Patients within this arm who have urine output <1 ml/kg/hr over 16 hours after the first dose of Lasix will be considered poor responders. These patients may be started on PD if clinically indicated. Those who show good response (urine output >1 ml/kg/hr over subsequent 16 hours) will continue furosemide as needed to augment urine output. If they subsequently develop oliguria or fluid overload unresponsive to diuretic therapy, these patients may later be started on PD at discretion of CICU attending with consultation of nephrology service.
  Interventions: Drug: Furosemide
- Peritoneal dialysis (Experimental): Patients within the PD arm will begin PD with a standardized dialysis plan of 10ml/kg of 1.5% Dianeal™ with 1 hours cycles (5 minute fill, 45 minute dwell and 10 minute drain). Further PD management will be directed by CICU attending and Nephrology service
  Interventions: Procedure: Peritoneal Dialysis

INTERVENTIONS:
Drug: Furosemide — Patients randomized to the furosemide arm will be given 1 mg/kg intravenously every 6 hours for 2 doses and then as directed by CICU attending to augment urine output. Patients within this arm who have urine output <1 ml/kg/hr over 16 hours after the first dose of Lasix will be considered poor responders. These patients may be started on PD if clinically indicated. Those who show good response (urine output >1 ml/kg/hr over subsequent 16 hours) will continue furosemide as needed to augment urine output. If they subsequently develop oliguria or fluid overload unresponsive to diuretic therapy, these patients may later be started on PD at discretion of CICU attending with consultation of nephrology service.
  Other Names: Lasix
  Arms: Furosemide
Procedure: Peritoneal Dialysis — Patients within the PD arm will begin PD with a standardized dialysis plan of 10ml/kg of 1.5% Dianeal™ with 1 hours cycles (5 minute fill, 45 minute dwell and 10 minute drain). Further PD management and discontinuation will be directed by CICU attending and Nephrology service.
  Other Names: PD
  Arms: Peritoneal dialysis

SUMMARY:
Acute kidney injury (AKI) after cardiopulmonary bypass (CPB) in infants is common and associated with poor outcomes. Peritoneal dialysis (PD) and furosemide have been used to attain negative fluid balance due to AKI induced oliguria, but have not been compared prospectively. The investigators will prospectively compare outcomes of infants with oliguria after CPB randomized to PD vs. furosemide with the hypothesis that infants receiving PD have superior outcomes.

DETAILED DESCRIPTION:
Background: Acute kidney injury (AKI) is a common postoperative complication after heart surgery with cardiopulmonary bypass (CPB). Multiple studies have demonstrated that patients with AKI have worse clinical outcomes, such as longer ventilation times and increased length of stay, which is thought to be secondary to associated oliguria and subsequent fluid overload. Studies suggest that early renal replacement therapy (RRT) via peritoneal dialysis (PD) may prevent fluid overload and therefore be a superior management to diuretic (i.e. furosemide) administration. However, there is no published evidence to suggest superiority or laboratory data available to guide decision making.

Objective: Our primary objective is to determine if early institution of PD improves clinical outcomes compared to administration of furosemide in post-operative cardiac infants with acute kidney injury. We hypothesize that early initiation of PD will improve clinical outcomes. We will determine if these clinical outcomes will be better among good responders of furosemide compared to poor responders. We will determine if postoperative NGAL concentrations are predictive of poor response to furosemide.

Design / Methods: The study will be a single-center randomized clinical trial among neonates undergoing cardiac surgery with CPB with planned placement of a PD catheter due to risk of AKI. If patients demonstrate oliguria within the first postoperative day, they will be randomized to early PD or trial of furosemide. Clinical and laboratory data will be collected and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 6 months of age;
* Undergoing cardiothoracic surgery with CPB;
* Planned placement of PD catheter per institutional standard of care criteria.

Exclusion Criteria:

* Pre-existing chronic kidney disease stage 3 or above (correlating with estimated GFR<60 ml/min/m2, which will be calculated using routine preoperative serum creatinine value using the modified Schwartz equation).
* Known history of allergy to furosemide.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Kwiatkowski, MD, Principal Investigator — Cinncinnati Children's Hospital Medical Center; Catherine D Krawczeski, MD, Study Director — Cinncinnati Children's Hospital Medical Center; Stuart L Goldstein, MD, Study Director — Cinncinnati Children's Hospital Medical Center
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data would be available to other researchers after publication of data at the discretion of the research team after communication with the PI

REFERENCES:
- [Derived] Kwiatkowski DM, Goldstein SL, Cooper DS, Nelson DP, Morales DL, Krawczeski CD. Peritoneal Dialysis vs Furosemide for Prevention of Fluid Overload in Infants After Cardiac Surgery: A Randomized Clinical Trial. JAMA Pediatr. 2017 Apr 1;171(4):357-364. doi: 10.1001/jamapediatrics.2016.4538. PMID 28241247
- See also: Center for Acute Care Nephology at Cincinnati Childrens — http://www.cincinnatichildrens.org/service/c/cacn/default/

RESULTS

PARTICIPANT FLOW:
Groups:
- Furosemide: Patients randomized to the furosemide arm will be given 1 mg/kg intravenously every 6 hours for 2 doses and then as directed by CICU attending to augment urine output. Patients within this arm who have urine output <1 ml/kg/hr over 16 hours after the first dose of Lasix will be considered poor responders. These patients may be started on PD if clinically indicated. Those who show good response (urine output >1 ml/kg/hr over subsequent 16 hours) will continue furosemide as needed to augment urine output. If they subsequently develop oliguria or fluid overload unresponsive to diuretic therapy, these patients may later be started on PD at discretion of CICU attending with consultation of nephrology service.
  Furosemide: Patients randomized to the furosemide arm are given 1 mg/kg intravenously every 6 hours for 2 doses and then as directed by CICU attending to augment urine output. Patients within this arm who have urine output <1 ml/kg/hr over 16 hours after the first dose of Lasix
- Peritoneal Dialysis: Patients within the PD arm will begin PD with a standardized dialysis plan of 10ml/kg of 1.5% Dianeal™ with 1 hours cycles (5 minute fill, 45 minute dwell and 10 minute drain). Further PD management will be directed by CICU attending and Nephrology service
  Peritoneal Dialysis: Patients within the PD arm will begin PD with a standardized dialysis plan of 10ml/kg of 1.5% Dianeal™ with 1 hours cycles (5 minute fill, 45 minute dwell and 10 minute drain). Further PD management and discontinuation will be directed by CICU attending and Nephrology service.
  One potential outcome during use of a peritoneal dialysis catheter is the development of a Pleural Peritoneal communication. In this event, dialysis fluid is instilled in the peritoneum and then leaks into the pleural space through a defect in the diaphragm. This fluid is then drained out of a surgical chest tube. This impairs the ability to perform peritoneal dialysis and thus is a reason to not complete the randomized arm.
Period: Overall Study
Arm/Group | Furosemide | Peritoneal Dialysis
Started | 32 | 41
Completed | 31 | 32
Not Completed | 1 | 9
Not completed — Physician Decision | 1 | 0
Not completed — Pleural Peritoneal communication | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Furosemide: Patients randomized to receive furosemide
- Peritoneal Dialysis: Patients randomized to receive peritoneal dialysis
- Total: Total of all reporting groups
Arm/Group | Furosemide | Peritoneal Dialysis | Total
Number analyzed (Participants) | 32 | 41 | 73
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 9 [7 to 14] | 8 [6 to 15] | 8 [6 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 21 | 26 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 31 | 40 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 29 | 37 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 32 | 41 | 73
Weight (kg) [Median (Inter-Quartile Range); unit: kg] | 3.4 [3 to 3.8] | 3.4 [3 to 3.8] | 3.4 [3 to 3.8]
Length (cm) [Median (Inter-Quartile Range); unit: cm] | 50 [47 to 53] | 50 [47 to 52] | 50 [47 to 52]
Baseline Creatinine (mg/dL) [Median (Inter-Quartile Range); unit: mg/dl] | 0.4 [0.36 to 0.5] | 0.4 [0.34 to 0.53] | 0.4 [0.34 to 0.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Negative Fluid Balance on Postop Day 1
Description: Difference of inputs and outputs, including urine output and PD drainage.
Time Frame: Postop day 1
Measure: Count of Participants; unit: Participants
Groups:
- Furosemide: Patients randomized to furosemide
- Peritoneal Dialysis: Patients randomized to peritoneal dialysis
Arm/Group | Furosemide | Peritoneal Dialysis
Number analyzed (Participants) | 32 | 41
Participants | 21 | 29

2. Secondary Outcome: Respiratory Support Administered
Description: Duration of initial course of postoperative mechanical ventilation
Time Frame: Duration of postoperative intubation (average time approximately- 1 week)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Furosemide | Peritoneal Dialysis
Number analyzed (Participants) | 32 | 41
days | 4 [2 to 6] | 3 [2 to 4]

3. Secondary Outcome: NGAL Concentration
Time Frame: Pre-op, and postop (2hr, 6hr, 12hr, 24hr, 48hr)
Population: Data were collected but not analyzed. Due to a high incidence of volatile and un-reportable NGAL levels, concerns were raised about the storage or processing of samples affecting data validity. Given the overwhelming concern of erroneous data, analysis was not performed as planned.
Groups:
- Peritoneal Dialysis: Patients randomized to PD
Arm/Group | Furosemide | Peritoneal Dialysis
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Cardiac ICU Stay
Description: Total days of initial postoperative stay in cardiac ICU
Time Frame: Average 2 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Furosemide | Peritoneal Dialysis
Number analyzed (Participants) | 32 | 41
days | 9 [5 to 15] | 7 [6 to 12]

5. Secondary Outcome: Duration of Hospital Stay
Description: Total days of initial postoperative stay in hospital
Time Frame: Average 4 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Furosemide | Peritoneal Dialysis
Number analyzed (Participants) | 32 | 41
days | 15 [10 to 28] | 14 [9 to 22]

6. Secondary Outcome: All Cause Mortality
Description: In-hospital mortality
Time Frame: duration of hospitalization (an average of 2 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide | Peritoneal Dialysis
Number analyzed (Participants) | 32 | 41
Participants | 3 | 1

7. Secondary Outcome: Renal/Electrolyte Abnormalities
Description: Total sum of renal and electrolyte abnormalities over the first 5 postoperative days as defined in the protocol
Time Frame: Postop morning 1-5
Measure: Median (Inter-Quartile Range); unit: abnormalities
Arm/Group | Furosemide | Peritoneal Dialysis
Number analyzed (Participants) | 32 | 41
abnormalities | 6 [4 to 7] | 4 [3 to 5]

8. Secondary Outcome: Doses of Potassium Chloride or Arginine Chloride Required
Description: Total doses of potassium chloride or arginine chloride given during the first five postoperative days.
Time Frame: Postop day 0-5
Measure: Median (Inter-Quartile Range); unit: doses given
Arm/Group | Furosemide | Peritoneal Dialysis
Number analyzed (Participants) | 32 | 41
doses given | 2 [1 to 5] | 1 [0 to 3]

9. Secondary Outcome: B-Natriuretic Peptide
Description: BNP measured at 24 and 48 hours postoperatively
Time Frame: At 24hours and 48 hours postoperative
Measure: Mean (Inter-Quartile Range); unit: pg/ml
Arm/Group | Furosemide | Peritoneal Dialysis
Number analyzed (Participants) | 32 | 41
pg/ml
  24 hours | 1334 [901 to 2764] | 1168 [555 to 2439]
  48 hours | 1110 [611 to 2221] | 663 [486 to 1593]

10. Secondary Outcome: Modified Oxygenation Index
Description: Product of Mean airway pressure delivered by mechanical ventilation and FiO2 of administered oxygen
Time Frame: at 24 and 48 hours postoperative
Measure: Median (Inter-Quartile Range); unit: Units
Arm/Group | Furosemide | Peritoneal Dialysis
Number analyzed (Participants) | 32 | 41
Units
  24 Hours | 4 [3.2 to 5.2] | 4 [0.03 to 5.4]
  48 Hours | 3.8 [2.4 to 5.4] | 2.8 [2.2 to 4.6]

ADVERSE EVENTS:
Arm/Group | Furosemide | Peritoneal Dialysis
All-Cause Mortality (participants affected / at risk) | 3/32 | 1/41
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/41
Other Adverse Events (participants affected / at risk) | 0/32 | 2/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Furosemide (N=32) | Peritoneal Dialysis (N=41)
Bleeding Event (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Bleeding from PD catheter or relating to its placement requiring blood product transfusion.
Hydrocele (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Development of hydrocele

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No